CLINICAL TRIAL: NCT04277130
Title: Intervention Study of Active Video Games on Intellectual Disabled Children's Physical Activity Level, Motor Ability and Physical Fitness
Brief Title: Effectiveness of Active Video Games in Children With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Lau Wing Chung, Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HASC/15-16/0169
Record Dates: First submitted 2020-02-12; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Intellectual Disability
Keywords: exergame; children with intellectual disability; physical activity; motor proficiency
MeSH Terms: conditions — Intellectual Disability; Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention with active video games
  Interventions: Behavioral: Intervention with active video games
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Intervention with active video games — Participants in intervention group were paired up by their teachers. Each participant had a classmate playing with him/her, and the waiting time is minimal because Xbox 360 Kinect allowed double play mode. The intervention group was provided with an AVG, the Xbox 360 Kinect technology (Kinect Sports Seasons I & II, including bowling, soccer, boxing, track and field, table tennis, beach volleyball, golf, tennis). The AVG intervention consisted of two 30-min sessions per week, for a total of 12 weeks. Participants either played in PE classes and/or recess. They had no other specific routing of activities but straight played the AVG during the intervention. They could free to choose games they like in the Xbox 360. The AVGs of Xbox 360 chosen was of moderate to vigorous intensity (3-6 METs) and no matter what games they chose, their PA level would be between moderate and vigorous intensity.
  Arms: Intervention group

SUMMARY:
Background: Children with intellectual disabilities (ID) are more vulnerable to obesity when compared to the normal children (Getchell et al., 2012; Maiano, 2011). Active video games (AVGs) on physical activity (PA) behavior have attracted academic interest and exploration since 2000. It has been demonstrated that an intervention with AVGs is compatible with the school setting and behavioral change in health and PA (Lau, et al., 2015). However, special populations such as ID children and their needs have been neglected in this area (Martins, Carvalho & Soares, 2011). ID children's PA behavior, motor ability and physical fitness is still an under-explored area.

Aims: To determine the effect of a prescribed AVG intervention on ID children's PA levels (sedentary, light, moderate, and vigorous), motor ability, and physical fitness. The intervention effects in children with mild intellectual disability will be explored.

Design: A standard two-arm parallel, single-blinded, randomized control cluster trial.

Schools: Participants will be recruited from six special schools in Hong Kong. Schools with same intellectual disability categories will be randomly assigned into intervention group and control group.

Participants: 200 Children aged 8~18 years old with intellectual disabilities will be recruited.

Intervention: ID children randomized to the intervention group will participate in an AVG intervention 60 minutes per week for 12 weeks in their PE class, in addition to their usual activity levels. The research team will prescribe updated AVG consistent with moderate-vigorous intensity.

Control: The control group will continue with usual PA alone and will not receive the AVG intervention.

Analysis: Repeated measures mixed model (2 groups X 2 time points (12-week post- test and 8-week follow up test)) by SPSS 23.0 will be used to investigate the intervention effect on primary and secondary outcomes, adjusting for baseline characteristics and correlation between repeated observations.

Significance: This will be the pioneering study to provide definitive evidence for the impact of a prescribed AVG intervention on ID children's PA level, motor ability and physical fitness. If effective, this research will provide significant evidence from the innovative method to inform health professionals and PE teachers how to incorporate AVG to enhance physical active behaviors, motor ability and physical fitness in ID children. Finally they may be able to enjoy a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* students with ID (mild category) aged 8-18 years old from special education schools including primary and secondary schools;

Exclusion Criteria:

* students without physical disability.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 203 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change of body mass index | through study completion, 12 weeks
  Weight (measured in kilograms) and height (measured in meters) are combined to report body mass index in kg/m^2. Change of body mass index between baseline and post-intervention test is assessed.
Change of body fat percentage | through study completion, 12 weeks
  Body fat percentage is measured using the Tanita BC-418 Body Composition Analyzer at baseline and post-intervention test and is reported the unit as %. Change of body fat percentage between baseline and post-intervention test is assessed.
Change of sedentary behavior time | through study completion, 12 weeks
  Objective physical activity level was recorded and measured using the ActiGraph GT3X+ activity monitor (Pensacola, FL). Counts per minute are recorded. The activity with lower than 100 counts per minute is categorized as sedentary behaviors. Overall time in sedentary behavior in minute is recorded as sedentary behavior time. Change of sedentary behavior time between baseline and post-intervention tests is assessed.
Change of light physical activity time | through study completion, 12 weeks
  Objective physical activity level was recorded and measured using the ActiGraph GT3X+ activity monitor (Pensacola, FL). Counts per minute are recorded. The activity with higher than 100 counts per minute but lower than 2296 counts per minute is categorized as light physical activity. Overall time in light physical activity in minute is recorded as light physical activity time. Change of light physical activity time between baseline and post-intervention tests is assessed.
Change of moderate-to-vigorous physical activity time | through study completion, 12 weeks
  Objective physical activity level was recorded and measured using the ActiGraph GT3X+ activity monitor (Pensacola, FL). Counts per minute are recorded. The activity with higher than 2296 counts per minute is categorized as moderate-to-vigorous physical activity. Overall time in moderate-to-vigorous physical activity in minute is recorded as moderate-to-vigorous physical activity time. Change of moderate-to-vigorous physical activity time between baseline and post-intervention tests is assessed.
Change of motor proficiency | through study completion, 12 weeks
  The short-form Bruininks-Oseretsky Test of Motor Proficiency™ - Second Edition (BOT-2) (Bruininks & Bruininks, 2005) is used for the assessment of motor proficiency. The scale consists of 14 items and scored 0-88. Higher score indicates higher motor proficiency. Change of BOT-2 score between baseline and post-intervention tests is assessed.
Change of muscular strength | through study completion, 12 weeks
  The hand dynamometer (Model 01160, Lafayette Instrument Company, Lafayette, Indiana, USA) is used to measure the muscular strength. Output is in kilograms (range 0.0-199.9kg with sensitivity at 0.1kg). The change of muscular strength between baseline and post-intervention tests is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Wing-Chung Lau, Ph.D, Principal Investigator — Hong Kong Baptist University

IPD SHARING:
Plan to Share IPD: No